CLINICAL TRIAL: NCT07110051
Title: Comparative Study Between Nalbuphine Versus Tramadol on Post Operative Analgesia in Abdominal Surgery on Pediatric Cancer Patient
Brief Title: Nalbuphine Versus Tramadol on Post Operative Analgesia in Abdominal Surgery on Pediatric Cancer Patient
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Norma Osama Abdalla Zayed, Lecturer of Anesthesia, Surgical ICU and Pain Management, National Cancer Institute, Cairo University, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AP2403-301-015
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Tramadol; Nalbuphine; Abdominal Surgeries; Pediatric Cancer
MeSH Terms: conditions — Neoplasms | interventions — Nalbuphine; Tramadol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nalbuphine (group A) (Active Comparator): group A (nalbuphine) will receive a single dose of nalbuphine (0.2 mg/kg) immediately after surgery to be repeated every 8 hours for the duration of the study (72 hours)
  Interventions: Drug: Nalbuphine
- Tramadol (group B) (Active Comparator): group B( Tramadol) will receive a single dose of tramadol (2 mg/kg) immediately after surgery to be repeated every 8 hours for the duration of the study (72 hours).
  Interventions: Drug: Tramadol

INTERVENTIONS:
Drug: Nalbuphine — this group will a single dose of nalbuphine (0.2 mg/kg) immediately after surgery to be repeated every 8 hours for the duration of the study (72 hours)
  Other Names: nalufin
  Arms: nalbuphine (group A)
Drug: Tramadol — this group will receive a single dose of tramadol (2 mg/kg) immediately after surgery to be repeated every 8 hours for the duration of the study (72 hours).
  Other Names: tramal
  Arms: Tramadol (group B)

SUMMARY:
In current study the investigators aim to compare between nalbuphine versus tramadol for post-operative pain control in abdominal surgeries in pediatric.

DETAILED DESCRIPTION:
Pain is an important and complex protective phenomenon. Good postoperative pain relief is important as it alleviates patient distress and aids a rapid, uncomplicated recovery.

Nalbuphine is a semi-synthetic opioid analgesic that belongs to the phenanthrene family. It is commonly used for pain management in children, but is associated with certain side effects such as respiratory and central nervous system depression, emesis, and pruritus due to its effect on µ2 receptors. Tramadol is a potent analgesic that binds to µ1 and µ2 receptors and enhances the inhibitory action of descending pain pathways. In contrast to other opioids, including nalbuphine, tramadol does not induce tolerance and is associated with reduced adverse effects.

Therefore, in this study, investigators will compare the efficacy of nalbuphine and tramadol for the management of postoperative pain in cancer children after abdominal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be children aged 3-12 years
* American society of anesthesia (ASA) classification I-III.
* scheduled for elective Abdominal surgery under general anesthesia

Exclusion Criteria:

* child guardian refusal.
* Allergy from Tramal or nalbuphine
* Patient with previous chronic pain on opioids

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
time to first rescue analgesia | 72 hours
  Time to first analgesic request( paracetamol)

SECONDARY OUTCOMES:
Frequency of paracetamol consumption | 72 hours
  Postoperative paracetamol frequency
Wong-barker faces pain rating scale score | 72 hours
  Wong-barker faces pain rating scale score will be measured every 8 hours. The Wong-Baker Faces Pain Rating Scale is a tool that uses a combination of faces, numbers, and words to help a person effectively communicate the severity of their physical pain.
  The scale starts at 0 and ends at 10, with the numbers increasing in intervals of 2. Each number relates to both a face and a small descriptive phrase. It is flexible because if someone uses the numbers, they may not need the faces or the wording. The phrase relating to each numerical value is as follows:
  0: no hurt or pain, 2: it hurts a little bit,4: it hurts a little more ,6: it hurts even more,8: it hurts a whole lot 10: it hurts the worst

CONTACTS AND LOCATIONS:
Overall Officials: Reham mohamed gamal, MD, Principal Investigator — assistant professor
Locations (1):
- National cancer institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for 6 months
Supporting Information: Study Protocol
Time Frame: After the end of study for 6 months
Access Criteria: The data will be available upon a reasonable request from the corresponding author.